CLINICAL TRIAL: NCT06995157
Title: Characteristics of Human Papillomavirus (HPV) Infections and HPV Vaccine Attitudes Among Slovenian Women After the Introduction of HPV Vaccination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: MSD Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0120-240/2023/3
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer Screening; Vaccination Uptake

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taking HPV sample and offering HPV vaccination (Other)
  Interventions: Biological: Offering HPV vaccine

INTERVENTIONS:
Biological: Offering HPV vaccine — During regular cervical cancer prevention visit with the gynecologist, HPV vaccine will be offered to participants 35 years or younger.

SUMMARY:
Cervical cancer (CC), primarily caused by persistent infection with high-risk human papillomavirus (HPV) types, remains a significant public health issue. Despite the availability of prophylactic HPV vaccines and improved screening methods, vaccination coverage and uptake remain suboptimal in many countries, including Slovenia. In 2020, the WHO launched a global strategy to eliminate CC, emphasizing 90% HPV vaccination coverage among girls, 70% screening of women at key ages, and 90% treatment of identified cases by 2030.

The EVEN FASTER concept proposes that targeting a specific age group of women-those bridging unvaccinated and vaccinated cohorts-with simultaneous HPV screening and vaccination may significantly reduce HPV transmission. Swedish data support this, showing a 62-64% reduction in high-risk HPV infections following combined interventions in women aged 23-30.

In Slovenia, HPV vaccination has been available since 2006 for girls, and since 2021 for boys, with average uptake around 50%. However, no comparable model has been implemented or studied locally. This proposed clinical study will assess HPV vaccine acceptability among women in Slovenia, identify barriers to uptake, define an optimal target age group for intervention, and evaluate the effectiveness of offering concurrent screening and vaccination to accelerate CC prevention in this region.

Women will be invited to participate during their preventive gynecological examination within Slovenia's national cervical cancer screening program (ZORA). Inclusion criteria include regular cervical smears (CS) every 3 years following a previously normal result, first or second CS after entering the ZORA program, follow-up CS after abnormal cytology, non-neoplastic findings, or cervical procedures, and CS due to clinical indications. Exclusion criteria include pregnancy, menstruation, cervical or vaginal inflammation, other medical conditions preventing CS collection, prior hysterectomy, prior CS taken for this study, or known hypersensitivity to HPV vaccine components.

Eligible women will be invited by the attending gynecologist and nurse. After the exam, participants will complete an anonymous questionnaire covering demographics, screening history, vaccination status, and vaccine attitudes. Assistance will be provided if needed.

Women aged ≤35 who are unvaccinated will receive counseling on HPV vaccination, including benefits and risks. Those consenting will receive free vaccination with the nonavalent Gardasil®9 vaccine, following a three-dose schedule (0, 1-2, 6 months).

Around 500 women aged ≤35 are expected in this sub-group, with fewer than half anticipated to accept vaccination. Data will be anonymized and analyzed using SPSS (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* regular cervical smear (CS) every 3 years after a previously normal CS result, first CS at entry into the ZORA screening program, second CS one year after entering the ZORA screening program following a previously normal first CS, control CS after a pathological cytological result or after a non-neoplastic cytological result or after conization or laser vaporization of the cervix, and curative CS due to signs or pathological clinical findings

Exclusion Criteria:

* pregnancy at the time of the gynecological examination, menstrual bleeding at the time of the gynecological examination, inflammation of the vagina and/or cervix at the time of the gynecological examination, other medical and clinical conditions that prevent the taking of a CS, condition after hysterectomy, already taken CS for the purpose of the present study, and hypersensitivity to the active substances or any excipient of the HPV vaccine

Max Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
HPV vaccine uptake | 2 years
  We expect 50% of participants to opt for vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Občina Domžale, Slovenia

IPD SHARING:
Plan to Share IPD: Yes